CLINICAL TRIAL: NCT06476964
Title: Stratification of Cutaneous Squamous Cell Carcinomas According to Its Transcriptomic, Metabolic and Inflammatory Characteristics
Acronym: StratiKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2024/07
Record Dates: First submitted 2024-06-19; First posted 2024-06-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Skin Cancer
Keywords: Actinic keratosis,; Cutaneous squamous cell carcinoma; mitochondria; metabolism
MeSH Terms: conditions — Skin Neoplasms; Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients with actinic keratosis(AK) (Experimental)
  Interventions: Procedure: skin biopsies
- patients with squamous cell carcinoma in situ (in situ cSCC) (Experimental)
  Interventions: Procedure: skin biopsies
- patients with squamous cell carcinomas infiltrative (infiltrative cSCC) (Experimental)
  Interventions: Procedure: skin biopsies
- patient with invasive metastases (cSCC with cutaneous metastases) (Experimental)
  Interventions: Procedure: skin biopsies

INTERVENTIONS:
Procedure: skin biopsies — Additional punches of 3 mm from a skin lesion part of a skin biopsy performed as part of routine care, an additional (optional) biopsy of healthy skin

SUMMARY:
A collection of biological samples (skin) will be created to meet the objectives. Skin biopsies will be taken (excluding on face and fold), in accordance with standard practice.

DETAILED DESCRIPTION:
Skin cancers are the most common type of cancer in human. Among them, cutaneous squamous cell carcinomas (cSCCs) represent the 2nd most frequent, with an incidence that continues to grow (+300% between 1994 and 2006) in line with the ageing of the population and sun exposure habits. cSCCs is a multi-stage carcinogenesis model: the pre-cancerous lesion is actinic keratosis (AK), which can either regress or progressively evolve into cSCC in situ and then infiltrating, and in some patients into a metastatic stage, initially lymph node and then distant, life-threatening. cSCCs are classified as low-risk or high-risk according to clinical and histological criteria associated with the risk of recurrence and metastasis. However, there is currently no tool for predicting this risk for a given cSCC, particularly according to its genetic characteristics. Indeed, the high mutation rate makes it difficult to identify specific genetic profiles. Similarly, there is no tool to predict the potential for a precancerous lesion (AK) to regress or to develop into a cSCC. The aim of this study is to characterize the molecular and metabolic features as well as immunologic landscapes of precancerous AK and cSCCs in order to uncover epithelial and immune cell subpopulations supporting tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over,
* Patients with suspected AK, or cSCC lesions (in situ, infiltrating or metastatic),
* Patients able to sign a consent form,
* Patients affiliated to a French Social Security system.

Exclusion Criteria:

* Patients who have previously received systemic treatment (chemotherapy, immunotherapy),
* Patients with cSCC or AK localized on visible zone of the face or folds
* Patients under guardianship or guardianship,
* Patient not affiliated to a French Social Security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Relative abundance of metabolite and differential enzyme expression in tumor lesion versus healthy tissue | Day 1
  Evaluation of metabolic changes involved in cSCC progression
Percentages of individual immune cell populations among total tumor-infiltrating immune cells will be evaluated. | Day 1
  Characterization of the immune cells infiltrate Expression of multiple immune cell markers will be assessed in samples from different subtypes of cSCC by single cell RNA sequencing.

SECONDARY OUTCOMES:
percentage of samples in each category (AK, in situ, ...) that present differentiation features are assessed by immunostaining of loricrin, filaggrin, K10 | Day 1
  Evaluation of skin differentiation markers
percentage of samples expressing aggressive markers will be assessed by evaluating the proliferation index | Day 1
  Evaluation of cSCC aggressiveness markers with the percentage of samples expressing aggressive markers will be assessed by evaluating the proliferation index, degree of differentiation, invasion beyond subcutaneous fat, perineural invasion, vascular invasion level of infiltration following immunohistochemistry analyses on formalin-fixed paraffin-embedded tissue sections.
percentage of samples that are highly proliferative will be calculated by measuring the ability of colony formation (SRB Test) | Day 1
  Evaluation of cancer proliferative features on skin biopsies with percentage of samples that are highly proliferative will be calculated by measuring the ability of colony formation (SRB Test) and cell cycle progression (flow cytometer, western).

CONTACTS AND LOCATIONS:
Overall Officials: Marie BEYLOT-BARRY, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Hamid-Reza REZVANI, PhD, Study Chair — Bordeaux Institute of Oncology
Locations (1):
- University Hospital of Bordeaux - Department of Dermatology, Bordeaux, France